CLINICAL TRIAL: NCT03871725
Title: Sonodynamic Therapy Manipulates Atherosclerosis Regression Trial on Patients With Carotid Atherosclerotic Plaques
Brief Title: Sonodynamic Therapy in the Treatment of Carotid Atherosclerosis
Acronym: SMART-C
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Principal Investigator, Ye Tian, Professor, MD, PhD, First Affiliated Hospital of Harbin Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMART-C pilot
Record Dates: First submitted 2019-03-08; First posted 2019-03-12 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Carotid Atherosclerosis
MeSH Terms: conditions — Carotid Artery Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sonodynamic therapy(SDT) (Experimental): Sonodynamic therapy(SDT) treatment is the combination of sonosensitizer administration and target atherosclerotic lesions ultrasound exposure.
  Interventions: Combination Product: Sonodynamic therapy (SDT)

INTERVENTIONS:
Combination Product: Sonodynamic therapy (SDT) — Sinoporphyrin sodium (DVDMS) as sonosensitizer, is dissolved in 0.9% sodium solution for following skin test and intravenous injection. 0.01mg/ml DVDMS solution (0.1ml) is prepared for skin test followed by 0.04 mg/ml DVDMS solution intravenous injection (0.2mg/kg).The target atherosclerotic lesions are marked on the corresponding skin with ultrasound guidance and underwent ultrasound exposure after 4 hours incubation. The therapeutic ultrasonic transducer is fixed to the marked skin site for 15min of each lesion. Ultrasound parameters included intensity of 1.6W/cm2 for carotid lesions, resonance frequency: 1.0 MHz and duty factor: 30%.

SUMMARY:
Sonodynamic therapy (SDT) is a new treatment for carotid atherosclerotic plaque. The purpose of this study is to evaluate the safety and initial effectiveness of this technique.

DETAILED DESCRIPTION:
Carotid atherosclerotic plaque is an important cause of ischemic stroke. Treatments for patients with carotid plaque include lifestyle changes, medical management(such as control of hyperlipidemia, hypertension, and diabetes) and carotid revascularization(carotid endarterectomy or carotid artery stenting). Studies have suggested that plaque morphology and composition are important determinants of plaque stability, using serial MR imaging of the carotid artery allowed observation of changes in plaque composition. Contrast enhanced ultrasound (CEUS) is a well accepted technique for detection of intraplaque neovascularization(IPN) in carotid atherosclerotic disease. The purpose of this trial is to evaluate the safety and initial effectiveness of SDT. The SDT can induce macrophage elimination and inhibit matrix degradation, which will promote plaque lipid depletion, inflammation level decrease and changes in other plaque tissue components, leading to plaque stabilization and reduction.

ELIGIBILITY:
Inclusion Criteria:

* Age 18- 80 years
* Carotid artery with 30%~70% stenosis by ultrasound and plaque thickness>2.5mm
* Patients without transient ischemic attack, minor stroke or amaurosis fugax within 6 months
* Patients' LDL-c level below 100 mg/dL(2.6mmol/L), well-controlled blood pressure(systolic BP<140 and diastolic BP<90 under resting conditions) and diabetes(HbA1c<7%)
* Written informed consent

Exclusion Criteria:

* Non-atherosclerotic carotid artery stenosis
* Contraindication to MRI( uses pacemaker, has metallic implants, claustrophobia)
* Acute MI, acute coronary syndrome or stroke within 4 weeks prior to visit
* Severe cerebral artery stenosis, atrial fibrillation or MRI detected thrombosis that would cause stroke
* Previous significant adverse reaction to a statin
* Systemic disorders such as hepatic, renal, hematologic, and malignant disease
* Medical history that might limit the individual's ability to take trial treatments for the duration of the study
* Allergic to DVDMS or sonovue
* Diagnosis of porphyria
* Pregnant women and nursing mothers
* History of bilateral carotid endarterectomy or has immediate plans for carotid endarterectomy
* Patient who is attending other clinical trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-01-05 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Change in plaque MaxWT, as assessed by MRI | Measured at Baseline, 1, 3, 6, and 9 months
  The changes in plaque MaxWT (maximum wall thickness) as assessed by MRI.

SECONDARY OUTCOMES:
Change in IPH volume, as assessed by MRI | Measured at Baseline, 1, 3, 6, and 9 months
  The changes in intraplaque hemorrhage (IPH) volume as assessed by MRI.
Change in LRNC volume, as assessed by MRI | Measured at Baseline, 1, 3, 6, and 9 months
  The changes in LRNC (lipid-rich necrotic core) volume as assessed by MRI.
Change in plaque LM volume, as assessed by MRI | Measured at Baseline, 1, 3, 6, and 9 months
  The changes in LM (loose matrix) volume as assessed by MRI.
Change in calcification volume, as assessed by MRI | Measured at Baseline, 1, 3, 6, and 9 months
  The changes in calcification (CA) volume as assessed by MRI.
Change in plaque volume, as assessed by MRI | Measured at Baseline, 1, 3, 6, and 9 months
  The changes in plaque volume(mm3) as assessed by MRI
Change in MVE, as assessed by CEUS | Measured at Baseline, 1, 3, 6, and 9 months
  The changes in normalised maximal video-intensity enhancement (MVE) are calculated to quantify the density of IPN as assessed by CEUS.
MACCE | Measured at Baseline, 1, 3, 6, and 9 months
  incidence of major adverse cardiovascular and cerebrovascular events(MACCE)
Incidence of adverse events | Measured at Baseline, 1, 3, 6, and 9 months
  Allergic to sunshine,hepatic or renal dysfunction,thyroid dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: YE TIAN, Study Chair — First Affiliated Hospital of Harbin Medical University
Locations (1):
- The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang, China